CLINICAL TRIAL: NCT00689494
Title: Cervical Device Contraception
Brief Title: Cervical Device Contraception-2 (Nanopaz)
Acronym: NANOPAZ
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Baram Paz, Bnai Zion MC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BnaiZionMC-08-BP-003-CTIL
Record Dates: First submitted 2008-05-19; First posted 2008-06-03 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-06

CONDITIONS: Healthy
Keywords: Nanopaz device; Blood progesterone measure in using the device; Delivery progesterone; Progesterone levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Nanopaz contraception device — levonorgestrel and levonorgestrel device for cervical contraception-nantechnolgy method
  Other Names: levonorgestrel device for cervical contraception-nantechnolgy method

SUMMARY:
Measure blood progesterone by using cervical device contraception.

DETAILED DESCRIPTION:
A very small cervical device that releases small amount of progesterone 20 mcgm/day.

The target of the research is to measure blood progesterone by using the cervical device.

This small device delivers progesterone by nanotechnology method.

ELIGIBILITY:
Inclusion Criteria:

* 10 healthy women are candidate for hysterectomy

Exclusion Criteria:

* Women with neoplastic malignancy disease or thrombophylia

Ages: 1 Month to 2 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-12 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
blood progesterone measure in blood | one to two months